CLINICAL TRIAL: NCT04614324
Title: A Prospective, Open Label, Multi-Center Study Using the RhinAer Procedure for Treatment of Subjects Suffering With Chronic Rhinitis
Brief Title: A Study of RhinAer ARC Stylus for Treating Chronic Rhinitis (RELIEF)
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP1056
Record Dates: First submitted 2020-10-27; First posted 2020-11-04 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Intervention Model Description: Active treatment for all subject enrolling prospectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- RhinAer ARC Stylus Treatment (Experimental): The RhinAer procedure will be performed in the study clinic using the RhinAer Stylus and Aerin Console. The RhinAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency energy to tissue when connected to the Aerin Console radiofrequency generating device. Participants will have both nostrils treated in the portion of the nasal cavity mucosa overlying the region of the posterior nasal nerve.
  Interventions: Device: RhinAer ARC Stylus

INTERVENTIONS:
Device: RhinAer ARC Stylus — The RhinAer procedure incorporates use of the RhinAer Stylus (Model FG815), which is a cleared (FDA - K192471) disposable handheld device capable of delivering bipolar radiofrequency energy to tissue. RhinAer has CE Marking in EU. The Aerin Console (Model FG226) RF generator with temperature control capable of delivering very low doses of energy was cleared for use in the US (FDA - K162810) and has CE Marking in the EU (CE639608).

SUMMARY:
Post-market study to continue to evaluate the effectiveness of the RhinAer ARC Stylus for chronic rhinitis.

DETAILED DESCRIPTION:
Prospective, Open Label, Multicenter Study of the Aerin Medical RhinAer® ARC Stylus for Chronic Rhinitis to continue to evaluate the effectiveness of the RhinAer® ARC Stylus for treating the posterior nasal nerve area to improve symptoms in adults diagnosed with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years (inclusively).
2. Willing and able to provide informed consent.
3. Willing and able to comply with the subject-specific requirements outlined in the Study Protocol.
4. Seeking treatment for chronic rhinitis symptoms of at least 6 months duration and willing to undergo an office-based procedure.
5. Moderate to severe symptoms of rhinorrhea (rTNSS rating of 2 or 3 for rhinorrhea).
6. Mild to severe symptoms of nasal congestion (rTNSS rating of 1, 2 or 3 for congestion).
7. rTNSS ≥ 6.

Exclusion Criteria:

1. Anatomic obstructions that in the investigator's opinion limit access to the posterior nasal passage.
2. Altered anatomy of the posterior nose as a result of prior sinus or nasal surgery or injury.
3. Active nasal or sinus infection.
4. History of significant dry eye.
5. History of any of the following: chronic epistaxis, documented episodes of significant nose bleeds in the past 3 months, rhinitis medicamentosa, head or neck irradiation.
6. Have rhinitis symptoms only on a seasonal basis due to allergies.
7. Known or suspected allergies or contraindications to the anesthetic agents and/or antibiotic medications to be used during the study procedure session.
8. Known or suspected to be pregnant or is lactating.
9. Participating in another clinical research study.
10. Has any condition that predisposes to excessive bleeding.
11. Is taking anticoagulants (eg, warfarin, Plavix) or 325 mg aspirin that cannot be discontinued before the procedure.
12. Has previous procedure or surgery for chronic rhinitis.
13. Other medical conditions which in the opinion of the investigator would predispose the subject to poor wound healing, increased surgical risk, or poor compliance with the requirements of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (12):
  - Arizona Desert ENT Specialists, Goodyear, Arizona
  - Sacramento ENT, Roseville, California
  - University of California, San Francisco, San Francisco, California
  - ENT Associates of South Florida, Boca Raton, Florida
  - ENT and Allergy Associates of Florida, Port Saint Lucie, Florida
  - Florida ENT and Allergy, Tampa, Florida
  - Chicago Nasal and Sinus Center, Chicago, Illinois
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Baton Rouge General / Sinus and Nasal Specialists of Louisiana, Baton Rouge, Louisiana
  - Piedmont ENT Associates, Winston-Salem, North Carolina
  - Fort Worth ENT, Fort Worth, Texas
  - ENT and Allergy Associates of Texas, McKinney, Texas
- Germany (3):
  - HNO-ZENTRUM am Kudamm, Berlin
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Facharzt für Hals- Nasen- und Ohrenkrankheiten Allergologie Plastische Operationen, Göttingen

IPD SHARING:
Plan to Share IPD: No
No data collected will be shared with other researchers participating in the study

REFERENCES:
- [Result] Lee JT, Abbas GM, Charous DD, Cuevas M, Goktas O, Loftus PA, Nachlas NE, Toskala EM, Watkins JP, Brehmer D. Two-Year Outcomes After Radiofrequency Neurolysis of Posterior Nasal Nerve in Chronic Rhinitis. Laryngoscope. 2024 May;134(5):2077-2084. doi: 10.1002/lary.31120. Epub 2023 Nov 2. PMID 37916848
- [Result] Lee JT, Abbas GM, Charous DD, Cuevas PDMM, Goktas PDMO, Loftus PA, Nachlas NE, Toskala EM, Watkins JP, Brehmer PDMD. Clinical and Quality of Life Outcomes Following Temperature-Controlled Radiofrequency Neurolysis of the Posterior Nasal Nerve (RhinAer) for Treatment of Chronic Rhinitis. Am J Rhinol Allergy. 2022 Nov;36(6):747-754. doi: 10.1177/19458924221109987. Epub 2022 Jul 11. PMID 35818709
- [Result] Kohlfaerber T, Pieper M, Munter M, Holzhausen C, Ahrens M, Idel C, Bruchhage KL, Leichtle A, Konig P, Huttmann G, Schulz-Hildebrandt H. Dynamic microscopic optical coherence tomography to visualize the morphological and functional micro-anatomy of the airways. Biomed Opt Express. 2022 May 5;13(6):3211-3223. doi: 10.1364/BOE.456104. eCollection 2022 Jun 1. PMID 35781952
- [Result] Lee JT, Abbas GM, Charous DD, Cuevas M, Goktas O, Loftus PA, Nachlas NE, Toskala EM, Watkins JP, Brehmer D. Three-Year Outcomes After Temperature-Controlled Radiofrequency Ablation of the Posterior Nasal Nerve for Chronic Rhinitis. Am J Rhinol Allergy. 2025 Nov;39(6):398-409. doi: 10.1177/19458924251360889. Epub 2025 Aug 4. PMID 40760831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this trial occurred between 10/5/2020 and 5/12/21. This prospective single-arm study enrolled patients across 16 centers in the United States (13) and Germany (3). All sites were either medical clinics or academic medical centers.
Pre-assignment Details: There was no wash out or run in for this study
Groups:
- Treatment Arm: Open Label, Single Arm Study - All subjects meeting eligibility requirements receive the Rhinaer Procedure
Period: Overall Study
Arm/Group | Treatment Arm
Started | 129
3Month | 128
6 Month | 123
Completed (Subjects still in follow up) | 0
Not Completed | 129
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2
Not completed — Remaining in Follow up | 123

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 105
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 117
  More than one race | 0
  Unknown or Not Reported | 3
Body Mass Index [Count of Participants; unit: Participants] — BMI stands for Body Mass Index, which is a measure of body fatness based on weight and height. BMI is calculated by dividing weight in kilograms by the square of height in meters
  Participants
    Underweight (<18.5) kg/m^2 | 4
    Normal (18.5-<25) kg/m^2 | 47
    Overweight (25-<30) kg/m^2 | 46
    Obese (30 & greater) kg/m^2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of the Reflective Total Nasal Symptoms Score (rTNSS)
Description: The rTNSS (Total Nasal Symptom Score) is a brief questionnaire developed to assess the severity of symptoms in individuals with rhinitis, particularly allergic rhinitis
  The questionnaire consists of questions that evaluate the following 4 symptoms of Nasal Congestion, Runny Nose, Nasal Itching and Sneezing.
  Each symptom is rated on a 4-point scale from "0" (no symptoms), "1" (mild symptoms), "2" (moderate symptoms" and "3" (severe symptoms). The total score is calculated by summing up the individual scores for each symptom.
  The total score is the sum of the 4 nasal symptoms.
  A low score indicates lower symptoms, a higher score indicates more symptoms. Range of score is 0-12 This questionnaire was provided to subjects at baseline and again at 3 months post procedure. This outcome measure shows the difference in overall scores. The average change in the score between baseline and 3M
Time Frame: Baseline and 3 months post study procedure
Measure: Mean (95% Confidence Interval); unit: Change in rTNSS score from baseline
Arm/Group | Treatment Arm
Number analyzed (Participants) | 128
Change in rTNSS score from baseline | -4.2 [-4.6 to -3.7]

2. Secondary Outcome: Participant Responder Percentage
Description: The rTNSS (Total Nasal Symptom Score) is a brief questionnaire developed to assess the severity of symptoms in individuals with rhinitis, particularly allergic rhinitis
  The questionnaire consists of questions that evaluate the following symptoms of Nasal Congestion, Runny Nose, Nasal Itching and Sneezing.
  Each symptom is rated on a 4-point scale from "0" (no symptoms) to "3" (severe symptoms). The total score is calculated by summing up the individual scores for each symptom.
  The total score is the sum of the 4 nasal symptoms.
  A low score indicates lower symptoms, a higher score indicates more symptoms. This questionnaire was provided to subjects at baseline and again at 3 months post procedure. This outcome measure shows the percentage of participants who responded to the procedure with improved rTNSS score
Time Frame: Baseline and 3 months post study procedure
Population: patients with an rTNSS at baseline and 3 months post procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RhinAer ARC Stylus Treatment
Number analyzed (Participants) | 126
percentage of participants | 76.2 [68.1 to 82.8]

3. Secondary Outcome: 3 Month - Mean Change in Mini Rhinoconjuctivitis Quality of Life Questionnaire (Mini RQLQ)
Description: The Rhinoconjuctivitis Quality of Life Questionnaire is validated rhinoconjuctivitis disease-specific instrument. The MiniRQLQ, to be used in this study, was developed and validated for efficiency by reducing the number of questions to 14.
  The instrument consists of 14 questions across 5 domains (activity limitations (n=3), practical problems (n=2), nose symptoms (n=3), eye symptoms (n=3), and other symptoms (n=3)). Responses are based on a 1-week recall and provided on a 7-point scale:
  * 0 = not troubled
  * 1 = hardly troubled at all
  * 2 = somewhat troubled
  * 3 = moderately troubled
  * 4 = quite a bit troubled
  * 5 = very troubled
  * 6 = extremely troubled.
  The total or overall MiniRQLQ score is the mean of the 14 responses (range of 0-6). Developers of the original RQLQ reported MCID for overall miniRQLQ >0.7 with another study indicating 0.42 (95% CI 0.30-0.51).
Time Frame: Baseline and 3 months post study procedure
Population: 127 subjects with MiniRQLQ scores at baseline and 3 months post treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 127
score on a scale | -1.8 [-1.8 to -1.4]

4. Secondary Outcome: 6 Months - Mean Change in Mini Rhinoconjuctivitis Quality of Life Questionnaire (Mini RQLQ)
Description: The Rhinoconjuctivitis Quality of Life Questionnaire is a well-established, validated, and the most frequently used rhinoconjuctivitis disease-specific instrument. The MiniRQLQ, to be used in this study, was developed and validated to further facilitate ease of use and efficiency by reducing the number of questions to 14.
  The instrument consists of 14 questions across 5 domains (activity limitations (n=3), practical problems (n=2), nose symptoms (n=3), eye symptoms (n=3), and other symptoms (n=3)). Responses are based on a 1-week recall and provided on a 7-point scale:
  * 0 = not troubled
  * 1 = hardly troubled at all
  * 2 = somewhat troubled
  * 3 = moderately troubled
  * 4 = quite a bit troubled
  * 5 = very troubled
  * 6 = extremely troubled.
  The total or overall MiniRQLQ score is the mean of the 14 responses range (0-6).
Time Frame: 6 Months
Population: Enrolled Subjects continuing at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 123
score on a scale | 1.17 (1.0)

5. Secondary Outcome: Number of Participants With Device Related Adverse Events
Description: Evaluate profile by characterizing the type and frequency of adverse events reported at or following the study procedure an throughout the follow up period
Time Frame: Baseline and 3 months post study procedure
Population: # of subjects experienced Device Related Adverse Event at 3months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 128
Participants | 0

6. Secondary Outcome: rTNSS Scores at 3 Months
Description: The TNSS is an instrument used to collect patient self-rated severity of nasal symptoms originally comprised of 3 symptoms (nasal obstruction, itching/sneezing and secretion/runny nose) that has been widely adapted to include 4 nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing. The patient rates 4 nasal symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing) on the following 4-point scale:
  * 0 = absent symptoms (no sign/symptom is evident)
  * 1 = mild symptoms (sign/symptom present, but minimal awareness; easily tolerated)
  * 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable)
  * 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping).
  The total score is the sum of the 4 nasal symptoms. Range of Scores 0-12
  A low score indicates lower symptoms, a higher score indicates more symptoms.
Time Frame: 3 Months
Population: Enrolled Subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 128
score on a scale | 3.56 (2.28)

7. Secondary Outcome: rTNSS Score at 6 Months
Description: as for outcome 6
Time Frame: 6 Months
Population: subjects treated and continuing on to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 123
score on a scale | 2.85 (2.24)

8. Secondary Outcome: rTNSS Change From Baseline at 6 Months Post Procedure
Description: as for outcome 6
Time Frame: 6 Months
Population: Subject continued on through 6 months. (3 lost to follow-up, 2 withdrew-consent, 1 withdrew by physician )
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 123
score on a scale | -4.90 (2.92)

ADVERSE EVENTS:
Time Frame: 3 years
Description: The definition for AE and SAE match Clinicaltrials.gov and follow ISO14144. Definitions also include Adverse Device Effect (ADE) ,Serious Adverse Device Effect (SADE), and unanticipated (Serious) Adverse Device Effect (UADE or USADE) based on (21 CFR 812.3)
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 0/129

LIMITATIONS AND CAVEATS:
Lack of a control arm and the limited follow-up to date It is possible that placebo effects may have contributed to the overall observed effect.

Medication use was not limited by the protocol Future research is needed to determine cost-benefit analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT04614324/Prot_SAP_000.pdf